CLINICAL TRIAL: NCT02315534
Title: A Phase Ib/II Clinical Study of BBI608 in Combination With Temozolomide for Adult Patients With Recurrent or Progressed Glioblastoma
Brief Title: A Study of BBI608 in Combination With Temozolomide in Adult Patients With Recurrent or Progressed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-251; BBI608-201GBM (Other: Boston Biomedical, Inc.)
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma
Keywords: GBM; Malignant Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — napabucasin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Patients for whom surgery is recommended as part of treatment for recurrent Glioblastoma.
  Interventions: Drug: BBI608; Drug: Temozolomide
- Arm B (Experimental): Patients for whom surgery is not recommended as part of the treatment for recurrent Glioblastoma.
  Interventions: Drug: BBI608; Drug: Temozolomide

INTERVENTIONS:
Drug: BBI608 — In arm A, BBI608 will be administered at the recommended Phase 2 dose (RP2D) twice daily for 7(±2) days prior to planned surgical resection or biopsy of recurrent GBM. Upon the clinical recovery of the patient and at a time between 15-28 days after surgery, BBI608 will be administered orally, daily, each day of a 28 day cycle in combination with temozolomide.
  In arm B, patients who are not candidates for surgical resection will receive BBI608 administered orally, daily, each day of a 28 day cycle at the RP2D in combination with temozolomide.
  Other Names: Napabucasin; BB608; BBI-608
Drug: Temozolomide — Temozolomide (TMZ) will be administered orally, once daily, at a dose of 150 mg/m^2 daily on days 1 through 5 of each 28-day study cycle. The dose of temozolomide can be increased to 200 mg/m^2 as per standard TMZ dosing guidelines for patients who complete at least one cycle at 150 mg/m^2.
  Other Names: Temodar

SUMMARY:
This is an open label, multi-center, phase 1 safety run-in and phase 2 study of BBI608 in combination with temozolomide in patients with recurrent or progressive glioblastoma who have not received prior bevacizumab therapy.

DETAILED DESCRIPTION:
In arm A, patients who are candidates for surgical resection will receive BBI608 as monotherapy prior to resection, followed by post-operative BBI608 administered in combination with temozolomide. In arm B, patients who are not candidates for surgical resection will receive BBI608 administered orally, daily, in combination with temozolomide.

In the phase 1/dose-limiting toxicity (DLT) cohort portion of this study, pharmacokinetics will be evaluated for both arms A and B. Pharmacodynamics will be evaluated in all patients who undergo surgical resection.

ELIGIBILITY:
Major Eligibility Criteria

1. Signed written informed consent must be obtained and documented according to International Conference on Harmonisation (ICH) and local regulatory requirements.
2. A histologically confirmed supratentorial glioblastoma (GBM) at first recurrence/progression (except for transformation from previous low grade glioma) following standard front-line therapy, for which treatment with temozolomide (TMZ) would be acceptable as determined by the Investigator
3. Previously received standard front-line GBM treatment including maximal surgical resection followed by external beam radiation therapy.
4. Patients may or may not be candidates for repeat surgical resection of the recurrent/progressed GBM.
5. Patients must have unequivocal evidence of tumor recurrence/progression by MRI at a minimum of 12 weeks following completion of chemoradiation or radiation therapy.
6. Patients must have measurable or non-measurable disease by response assessment in neuro-oncology Response Assessment in Neuro-oncology (RANO) criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03; Primary Completion 2018-10-09 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Laura and Isaac Perlmutter Cancer Center, New York, New York, United States
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are no pre-assignment details, study arm was determined at patient enrollment to the study
Groups:
- Candidates Whom Surgery is Recommended.: BBI608 will be administered at the recommended phase 2 dose (RP2D) twice daily for 7(±2) days prior to planned surgical resection or biopsy of recurrent GBM. Upon the clinical recovery of the patient and at a time between 15-28 days after surgery, BBI608 will be administered orally, daily, each day of a 28 day cycle in combination with temozolomide
- Candidates Whom Surgery is Not Recommended.: Patients who are not candidates for surgical resection will receive BBI608 administered orally, daily, each day of a 28 day cycle at the recommended phase 2 dose (RP2D) in combination with temozolomide
Period: Overall Study
Arm/Group | Candidates Whom Surgery is Recommended. | Candidates Whom Surgery is Not Recommended.
Started | 4 | 30
Assessment of Dose-limiting Toxicity (DLT) | 0 | 0
Off Treatment Due to Radiologic Disease Progression (PD) | 2 | 20
Off Treatment Due to Clinically Unacceptable Toxicities | 1 | 7
Off Treatment Due to Patient Request | 1 | 2
Off Treatment Due to Clinical PD | 0 | 1
Completed | 4 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Candidates Whom Surgery is Recommended.: Candidates who were candidates for repeat surgical resection
- Candidates Whom Surgery is Not Recommended: Candidates who were not candidates for repeat surgical resection
- Total: Total of all reporting groups
Arm/Group | Candidates Whom Surgery is Recommended. | Candidates Whom Surgery is Not Recommended | Total
Number analyzed (Participants) | 4 | 30 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (10.14) | 54.6 (15.54) | 55.1 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 12 | 14
  Male | 2 | 18 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 26 | 26
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 0 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking [Count of Participants; unit: Participants]
  Lifetime nonsmoker | 3 | 21 | 24
  Current smoker | 0 | 2 | 2
  Former smoker | 1 | 7 | 8
Weight [Mean (Standard Deviation); unit: kilograms] | 100.55 (26.345) | 78.21 (16.170) | 80.84 (13.608)
Height [Mean (Standard Deviation); unit: centimeters] | 177.25 (7.411) | 173.91 (9.896) | 174.30 (9.605)

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities (DLTs)
Description: Number of patients who experienced a dose limiting toxicity following a dosing of BBI608
Time Frame: 28 days after first administration of combination treatment (BBI608+TMZ)
Population: Up to the first 6 patients whom surgery was and wasn't recommended that received 28 days of continuous daily administration of BBI608 in combination with TMZ. Patients also had to be≥ 80% compliant to assigned dose to qualify for DLT analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Candidates Whom Surgery is Recommended.: The first 6 patients whom surgery was recommended that received 28 days of continuous daily administration of BBI608 in combination with TMZ. Patients also had to be ≥ 80% compliant to assigned dose to qualify for DLT analysis.
- Candidates Whom Surgery is Not Recommended: The first 6 patients whom surgery was not recommended that received 28 days of continuous daily administration of BBI608 in combination with TMZ. Patients also had to be ≥ 80% compliant to assigned dose to qualify for DLT analysis.
Arm/Group | Candidates Whom Surgery is Recommended. | Candidates Whom Surgery is Not Recommended
Number analyzed (Participants) | 4 | 6
Participants | 0 | 0

2. Primary Outcome: Progression Free Survival (PFS)-6
Description: To assess the effect of BBI608 + temozolomide (TMZ) therapy defined as the percentage of patients who have survived without objective disease progression for at least 6 months after treatment per neuro-oncology (RANO) criteria who had evaluable disease at baseline. PFS-6 is defined as the percentage of patients who survived without objective disease progression per RANO criteria for at least 6 months after treatment.
Time Frame: From the time of exposure to study drug to first objective documentation of disease progression or death due to any cause, assessed up to 6 months
Population: Data was only collected and analyzed for arms that enrolled at least 10 evaluable patients.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Candidates Whom Surgery is Not Recommended.: Participants who were not recommended for surgery that had evaluable disease at baseline and received at least 28 days of study drug (BBI608) in combination with temozolomide (TMZ). Data was only collected and analyzed for arms that enrolled at least 10 evaluable patients.
- Candidates Whom Surgery is Recommended.: Participants who were recommended for surgery that had evaluable disease at baseline and received at least 28 days of study drug (BBI608) in combination with temozolomide (TMZ). Data was only collected and analyzed for arms that enrolled at least 10 evaluable patients.
Arm/Group | Candidates Whom Surgery is Not Recommended. | Candidates Whom Surgery is Recommended.
Number analyzed (Participants) | 30 | 0
percentage of participants | 28.07 [16.81 to 40.45] |

3. Secondary Outcome: Progression Free Survival (PFS)-12
Description: To assess the effect of BBI608 + temozolomide (TMZ) therapy defined as the percentage of patients who have survived without objective disease progression for at least 12 months after treatment per neuro-oncology (RANO) criteria who had evaluable disease at baseline. PFS-12 is defined as the percentage of patients who survived without objective disease progression per RANO criteria for at least 12 months after treatment.
Time Frame: From the time of exposure to study drug to first objective documentation of disease progression or death due to any cause, up to 12 months
Population: Data was only collected and analyzed for arms that enrolled at least 10 evaluable patients.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Candidates Whom Surgery is Not Recommended | Candidates Whom Surgery is Recommended
Number analyzed (Participants) | 30 | 0
percentage of participants | 16.84 [7.84 to 28.75] |

4. Secondary Outcome: Overall Survival (OS)
Description: To assess the effect of BBI608 + temozolomide (TMZ) on the overall survival of patients with recurrent or progressive glioblastoma multiforme (GBM) who had not received prior treatment with bevacizumab or other anti-vascular endothelial growth factor agents who either were eligible or not eligible for surgical resection.
Time Frame: From the time of exposure to study drug to death from any cause. If patient discontinued study drug, they were assessed the first 3 months after discontinuation, then every 3 months up to 1 year, then every 6 months thereafter until death.
Population: Data was only collected and analyzed for arms that enrolled at least 10 evaluable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Candidates Whom Surgery is Not Recommended | Candidates Whom Surgery is Recommended
Number analyzed (Participants) | 30 | 0
months | 8.05 [6.01 to 10.87] |

5. Secondary Outcome: Disease Control Rate (DCR)
Description: To assess the percentage of patients that had evaluable disease at baseline with a documented complete response, partial response, and stable disease (CR + PR + SD) based on the Response Assessment in Neuro-Oncology (RANO) criteria out of all patients who received at least one dose of any study drug and had evaluable disease at baseline.
Time Frame: 4 weeks
Population: Data was only collected and analyzed for arms that enrolled at least 10 evaluable patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Candidates Whom Surgery is Not Recommended | Candidates Whom Surgery is Recommended
Number analyzed (Participants) | 30 | 0
percentage of patients | 30 [14.7 to 49.4] |

6. Secondary Outcome: Overall Response Rate (ORR)
Description: The proportion of patients with a documented complete response and partial response (CR + PR) based on RANO criteria.
Time Frame: 4 weeks
Population: Data was only collected and analyzed for arms that enrolled at least 10 evaluable patients.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Candidates Whom Surgery is Not Recommended | Candidates Whom Surgery is Recommended
Number analyzed (Participants) | 30 | 0
percentage | 3 [2.1 to 10.87] |

7. Secondary Outcome: Pharmacokinetic Profile of BBI608 and Temozolomide When Administered in Combination With Temozolomide as Assessed by the Area Under the Curve
Description: The area under the curve of BBI608, from time 0 to the last quantifiable concentration, calculated by a combination of linear and logarithmic trapezoidal methods (linear up/log down method)
Time Frame: On Day 1 and Day 5 after the first dosing, prior to dosing and 1, 2, 3, 5, 5h40m (day 1 only), 6, 7, 8 and 24 hours after first dose of BBI608
Population: Candidates for who surgery was and was not recommended that received at least one dose of study drug and had at least one quantifiable concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Groups:
- Candidates Whom Surgery is Recommended: Candidates whom surgery is recommended that received at least one dose of study drug and had at least one quantifiable concentration
- Candidates Whom Surgery is Not Recommended: Candidates for whom surgery was not recommended that received at least one dose of study drug and had at least one quantifiable concentration
Arm/Group | Candidates Whom Surgery is Recommended | Candidates Whom Surgery is Not Recommended
Number analyzed (Participants) | 4 | 10
h*ng/ml | 4820 (19) | 4200 (37.4)

8. Secondary Outcome: Pharmacodynamic Activity of BBI608 When Administered in Combination With Temozolomide as Assessed by Tumor Biopsy and Cancer Stem Cell Assays as Well as the Concentration of Study Drug in Tumors
Description: Tumor samples to provide information of the biomarkers by histopathology and Cancer Stem Cell assays as well as the concentration of study drug in tumors.
Time Frame: At the time of surgical resection
Population: Candidates whom surgery is either recommended or nor recommended that received 28 days of study drug and provided tissue samples.
Measure: Count of Participants; unit: Participants
Groups:
- Candidates Whom Surgery is Not Recommended; Candidates Whom Surgery is Recommended: Candidates whom surgery is either recommended or not recommended that received 28 days of study drug and provided tissue samples
Arm/Group | Candidates Whom Surgery is Not Recommended | Candidates Whom Surgery is Recommended
Number analyzed (Participants) | 23 | 0
Participants
  pSTAT3+ | 19 |
  pSTAT3- | 2 |
  Not Applicable | 2 |

ADVERSE EVENTS:
Time Frame: Every 1-2 weeks from study enrollment until end of treatment. Following last dose, follow-up period of 30 days.
Groups:
- Candidates Whom Surgery is Recommended: Participants whom surgery was recommended and received at least one dose of study medication (BBI608).
- Candidates Whom Surgery is Not Recommended: Patients who were not candidates for surgical resection and received at least one dose of study medication (BBI608).
Arm/Group | Candidates Whom Surgery is Recommended | Candidates Whom Surgery is Not Recommended
All-Cause Mortality (participants affected / at risk) | 4/4 | 22/30
Serious Adverse Events (participants affected / at risk) | 3/4 | 5/30
Other Adverse Events (participants affected / at risk) | 4/4 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candidates Whom Surgery is Recommended (N=4) | Candidates Whom Surgery is Not Recommended (N=30)
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candidates Whom Surgery is Recommended (N=4) | Candidates Whom Surgery is Not Recommended (N=30)
Diarrhoea (Gastrointestinal disorders) | 3 | 27
Abdominal pain (Gastrointestinal disorders) | 2 | 21
Nausea (Gastrointestinal disorders) | 1 | 14
Vomiting (Gastrointestinal disorders) | 1 | 10
Constipation (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 10
Pyramidal tract syndrome (Nervous system disorders) | 1 | 5
Aphasia (Nervous system disorders) | 2 | 4
Dysarthria (Nervous system disorders) | 0 | 4
Hemiparesis (Nervous system disorders) | 1 | 4
Cognitive disorder (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 3
Memory Impairment (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 3
Hemianopia homonymous (Nervous system disorders) | 1 | 2
Seizure (Nervous system disorders) | 1 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 2 | 0
Fatigue (General disorders) | 4 | 16
Gait disturbance (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 3 | 0
Lymphocyte count decreased (Investigations) | 0 | 6
Platelet count decreased (Investigations) | 1 | 6
Weight decreased (Investigations) | 1 | 5
Alanine aminotransferase increased (Investigations) | 1 | 4
Neutrophil count decreased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 2
Weight Increased (Investigations) | 0 | 2
White blood cell count decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 3 | 2
Chromaturia (Renal and urinary disorders) | 1 | 4
Hypotension (Vascular disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT02315534/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT02315534/SAP_001.pdf